CLINICAL TRIAL: NCT00874666
Title: Allicin Bioavailability of Garlic Products
Brief Title: Allicin Bioavailability From Garlic Supplements and Garlic Foods
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Silliker, Inc. (Industry)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Larry D. Lawson, principal investigator, Silliker, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: R21AT004236 (NIH); R21AT004236 (NIH); 1R21AT004236-01 (NIH)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: garlic; allicin; allyl methyl sulfide; healthy persons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Positive control with 100% allicin bioavailability
  Interventions: Other: crushed garlic clove
- 2 (Experimental): garlic powder tablet
  Interventions: Dietary Supplement: garlic powder tablet

INTERVENTIONS:
Other: crushed garlic clove — 1 gram crushed garlic in gelatin capsules, one dose once every 2-16 weeks
  Other Names: Allium sativum
  Arms: 1
Dietary Supplement: garlic powder tablet — tablets, dose to contain 1 gram of garlic powder, consume one dose once every two weeks for up to 52 weeks
  Other Names: Kwai, Garlique
  Arms: 2

SUMMARY:
This study will measure the bioavailability of allicin, the main active compound of garlic, from garlic supplements and garlic foods (raw, cooked, processed) so that

* supplement manufacturers and clinical investigators know how supplements need to be made and consumed to obtain high bioavailability
* consumers can know how garlic can be prepared to obtain any established health benefits of garlic.

DETAILED DESCRIPTION:
The bioavailability of allicin, the main active compound of garlic, from garlic supplements and garlic foods is highly questionable and unpredictable from in vitro tests, due to dependence upon alliinase activity under conditions that challenge alliinase activity (heat, gastric acid, intestinal proteases). It is likely that garlic supplement manufacturing procedures and coatings, meal conditions when supplements are consumed (high or low protein), and garlic food preparation conditions (temperature, surface area) will greatly affect allicin bioavailability. Such variability may account for some of the many conflicts seen in clinical trials on cardiovascular disease risk factors.

To resolve these issues, this study will determine the actual bioavailability of allicin from several types of garlic supplements and garlic foods under various conditions. Bioavailability will be determined by measuring the area under the 32-hour curve for breath concentrations of allyl methyl sulfide, the main metabolite allicin.

ELIGIBILITY:
Inclusion Criteria:

* in good health (self-judged)
* BMI (body mass index): 19-32 kg/m2
* not planning to move out of the area in the next year
* willing to abstain from consuming garlic and onion and foods that contain them for two days prior to and during each test (diet restrictions)
* able to deliver bags of breath to the research facility five times in two days
* willing to eat whole wheat tuna sandwiches

Exclusion Criteria:

* known serious health problems: diabetes, heart disease, active neoplasms, renal or liver disease, hyper- or hypothyroidism, breathing disorders, gastroesophageal reflux disease (GERD), gastrointestinal disease (absorption interference)
* known allergy to garlic or wheat
* tobacco user
* excessive alcohol intake (³2 drinks/day, self-reported)
* unable to speak English well

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Breath allyl methyl sulfide | 1-32 hours

CONTACTS AND LOCATIONS:
Overall Officials: Larry D Lawson, Ph. D., Principal Investigator — Silliker, Inc.
Locations (1):
- Silliker, Inc., Orem, Utah, United States